CLINICAL TRIAL: NCT06085807
Title: Using Culturally-sensitive Discussions and Genetic Testing to Improve Access to Early Autosomal Dominant Polycystic Kidney Disease Care and Improve Health Disparities
Brief Title: Genetic Testing in Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: P0568093
Record Dates: First submitted 2023-10-02; First posted 2023-10-17 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ADPKD: The participants will receive a survey.
  Interventions: Other: Survey
- Family members of patients with ADPKD: The family members of participants will receive a survey.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Groups will receive a survey to assess attitudes about diagnosis, treatment, and genetic testing in ADPKD.

SUMMARY:
Individuals with a diagnosis of autosomal dominant polycystic kidney disease (ADPKD) often have a family history of the condition although up to 10-15% of cases are sporadic mutations. The investigators recently conducted an analysis of the investigators clinic population to determine percentages of individuals who have undergone kidney imaging and genetic testing and determined total numbers of patients eligible for tolvaptan and those currently active on tolvaptan. The study team found large racial discrepancies in usage of tolvaptan and found that more patients are eligible for tolvaptan than are currently taking the medication. Reasons for this are often due to patient perception about the medication rather than treatment failure. There is a strong medical need to understand reasons for underuse of this critical medication in this population. Among those with genetic testing, the study team found large disparities in ethnic background between individuals offered genetic testing who accept versus decline testing. The study team also found that those who choose to pursue genetic testing are more likely to have no family history of the condition, presumably because the diagnosis is more "surprising" to them and thus desire for verification by genetic testing, if possible, is greater. However, it is known that genetic testing can be an important component of understanding of disease biology in all patients with ADPKD, while also providing important clinical information in some cases as individuals prepare for living donor transplantation or family planning. The investigators seek to understand barriers to use of tolvaptan and genetic testing among individuals in the clinic population and their relatives across a wide range of racial and ethnic backgrounds. The investigators hypothesize that anxiety about genetic conditions in particular is a barrier to accepting testing. The investigators seek to understand the mental health aspects of the diagnosis of ADPKD. They will also evaluate changes in symptoms compared to pre-treatment after initiation of tolvaptan in eligible individuals using qualitative techniques. In so doing, the study team hope to improve care for current patients and also to expand the pool of the clinic population to include newly diagnosed family members ideally at early stages of disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADPKD

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals affected by ADPKD and their family members
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Questionnaire responses regarding anxiety, genetics, and genetic testing attitudes in PKD participants and family members. | The investigators will administer one baseline survey over a recruitment time frame of 4 weeks and thereafter solicit family member participation for one-time survey measurements through study completion, up to one year.
  The survey incorporates the GAD4 questionnaire, which has scores graded from 0-3. It also includes questions graded on a Likert scale (1-5). The outcome measures will be reported as mean (SD) for each question on the survey.
  The investigators have developed a survey entitled "Anxiety, genetics, and polycystic kidney disease" incorporating elements of the GAD-4 questionnaire and tools developed by Lidewij Henneman to evaluate genetic testing attitudes among the general public.

CONTACTS AND LOCATIONS:
Overall Officials: Meyeon Park, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD not being shared.